CLINICAL TRIAL: NCT02519257
Title: The Relationship of Adiponectin in Adipose Tissue, Thy-1 in Plaques, and Inflammatory
Brief Title: The Relationship of Adiponectin in Adipose Tissue, Thy-1 in Plaques, and Inflammatory Mediators With Cardiac Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Shu-Hsun Chu, President, Far Eastern Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FEMH-96091
Record Dates: First submitted 2015-08-02; First posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Heart Surgery
Keywords: CAD; VHD; Thy-1
MeSH Terms: interventions — JCAD protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAD (Experimental): Patients with valve diseases proposed to have cardiac operations will be enrolled in this study, but those with congestive heart failure are excluded. Besides, those patients with valve diseases should have patent coronary arteries on coronary angiography.
  Interventions: Procedure: CAD
- VHD (Experimental): Patients with valve diseases proposed to have cardiac operations will be enrolled in this study, but those with congestive heart failure are excluded. Besides, those patients with valve diseases should have patent coronary arteries on coronary angiography.
  Interventions: Procedure: VHD

INTERVENTIONS:
Procedure: CAD — Patients with CAD diseases proposed to have cardiac operations will be enrolled in this study, but those with congestive heart failure are excluded. Besides, those patients with valve diseases should have patent coronary arteries on coronary angiography.
  Other Names: coronary artery disease
  Arms: CAD
Procedure: VHD — Patients with valve diseases proposed to have cardiac operations will be enrolled in this study, but those with congestive heart failure are excluded. Besides, those patients with valve diseases should have patent coronary arteries on coronary angiography.
  Other Names: valve diseases
  Arms: VHD

SUMMARY:
Atherosclerosis is an inflammatory process in which immune mechanisms interact with metabolic risk factors to initiate, propagate, and activate lesions in the arterial trees and is known as the main cause of coronary artery disease (CAD). Recently, there are more and more studies highlighted the potential importance of adipose tissue in relation to inflammation effects on CAD pathogenesis. However, it remains unclear whether Thy-1, adiponectin or any other inflammatory mediators in mediastinal adipose tissue contribute to CAD. In this study, we aim to analyze the expression of inflammatory mediators' expression via in vitro assay (3T3-L1 cell culture) and in vivo assay (human adipose tissues).

DETAILED DESCRIPTION:
In addition, we'd like to investigate the association of the investigators' findings with clinical atherosclerotic risks, medications (statins or antiplatelet), and blood sugar. Now, we've established cell assay and successfully transformed mature adipocyte from 3T3-L1 cells. Besides, there were nighty-six patients enrolled into this study. Flow cytometry of Thy-1 and MCP-1 concentration in cultured medium by ELISA were also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* coronary artery bypass grafting surgery
* valvular surgery

Exclusion Criteria:

* liver disease (GPT 2 times greater than normal limits)
* chronic renal insufficiency (Creatinine > 2.0 mg/dL)
* neoplastic diseases
* taking steroids
* congestive heart failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
CD91 (Thy-1) | up to 24 months

SECONDARY OUTCOMES:
CD45 | up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

REFERENCES:
- [Background] Lindahl B, Toss H, Siegbahn A, Venge P, Wallentin L. Markers of myocardial damage and inflammation in relation to long-term mortality in unstable coronary artery disease. FRISC Study Group. Fragmin during Instability in Coronary Artery Disease. N Engl J Med. 2000 Oct 19;343(16):1139-47. doi: 10.1056/NEJM200010193431602. PMID 11036119
- [Background] Ridker PM, Rifai N, Stampfer MJ, Hennekens CH. Plasma concentration of interleukin-6 and the risk of future myocardial infarction among apparently healthy men. Circulation. 2000 Apr 18;101(15):1767-72. doi: 10.1161/01.cir.101.15.1767. PMID 10769275
- [Background] Ridker PM, Rifai N, Pfeffer M, Sacks F, Lepage S, Braunwald E. Elevation of tumor necrosis factor-alpha and increased risk of recurrent coronary events after myocardial infarction. Circulation. 2000 May 9;101(18):2149-53. doi: 10.1161/01.cir.101.18.2149. PMID 10801754
- [Background] Shimokawa H, Ito A, Fukumoto Y, Kadokami T, Nakaike R, Sakata M, Takayanagi T, Egashira K, Takeshita A. Chronic treatment with interleukin-1 beta induces coronary intimal lesions and vasospastic responses in pigs in vivo. The role of platelet-derived growth factor. J Clin Invest. 1996 Feb 1;97(3):769-76. doi: 10.1172/JCI118476. PMID 8609234
- [Background] Miyata K, Shimokawa H, Kandabashi T, Higo T, Morishige K, Eto Y, Egashira K, Kaibuchi K, Takeshita A. Rho-kinase is involved in macrophage-mediated formation of coronary vascular lesions in pigs in vivo. Arterioscler Thromb Vasc Biol. 2000 Nov;20(11):2351-8. doi: 10.1161/01.atv.20.11.2351. PMID 11073837
- [Background] Mazurek T, Zhang L, Zalewski A, Mannion JD, Diehl JT, Arafat H, Sarov-Blat L, O'Brien S, Keiper EA, Johnson AG, Martin J, Goldstein BJ, Shi Y. Human epicardial adipose tissue is a source of inflammatory mediators. Circulation. 2003 Nov 18;108(20):2460-6. doi: 10.1161/01.CIR.0000099542.57313.C5. Epub 2003 Oct 27. PMID 14581396
- [Background] Prescott MF, McBride CK, Court M. Development of intimal lesions after leukocyte migration into the vascular wall. Am J Pathol. 1989 Nov;135(5):835-46. PMID 2817082
- [Background] Ouchi N, Kihara S, Arita Y, Maeda K, Kuriyama H, Okamoto Y, Hotta K, Nishida M, Takahashi M, Nakamura T, Yamashita S, Funahashi T, Matsuzawa Y. Novel modulator for endothelial adhesion molecules: adipocyte-derived plasma protein adiponectin. Circulation. 1999 Dec 21-28;100(25):2473-6. doi: 10.1161/01.cir.100.25.2473. PMID 10604883
- [Background] Staiger H, Tschritter O, Machann J, Thamer C, Fritsche A, Maerker E, Schick F, Haring HU, Stumvoll M. Relationship of serum adiponectin and leptin concentrations with body fat distribution in humans. Obes Res. 2003 Mar;11(3):368-72. doi: 10.1038/oby.2003.48. PMID 12634431
- [Background] Yatagai T, Nagasaka S, Taniguchi A, Fukushima M, Nakamura T, Kuroe A, Nakai Y, Ishibashi S. Hypoadiponectinemia is associated with visceral fat accumulation and insulin resistance in Japanese men with type 2 diabetes mellitus. Metabolism. 2003 Oct;52(10):1274-8. doi: 10.1016/s0026-0495(03)00195-1. PMID 14564678
- [Background] Matsuzawa Y. Adipocytokines and metabolic syndrome. Semin Vasc Med. 2005 Feb;5(1):34-9. doi: 10.1055/s-2005-871744. PMID 15968578
- [Background] Filippi E, Sentinelli F, Romeo S, Arca M, Berni A, Tiberti C, Verrienti A, Fanelli M, Fallarino M, Sorropago G, Baroni MG. The adiponectin gene SNP+276G>T associates with early-onset coronary artery disease and with lower levels of adiponectin in younger coronary artery disease patients (age <or=50 years). J Mol Med (Berl). 2005 Sep;83(9):711-9. doi: 10.1007/s00109-005-0667-z. Epub 2005 May 5. PMID 15877215
- [Background] Shimabukuro M, Higa N, Asahi T, Oshiro Y, Takasu N, Tagawa T, Ueda S, Shimomura I, Funahashi T, Matsuzawa Y. Hypoadiponectinemia is closely linked to endothelial dysfunction in man. J Clin Endocrinol Metab. 2003 Jul;88(7):3236-40. doi: 10.1210/jc.2002-021883. PMID 12843170
- [Background] Fernandez-Real JM, Lopez-Bermejo A, Casamitjana R, Ricart W. Novel interactions of adiponectin with the endocrine system and inflammatory parameters. J Clin Endocrinol Metab. 2003 Jun;88(6):2714-8. doi: 10.1210/jc.2002-021583. PMID 12788878
- [Background] Yokota T, Oritani K, Takahashi I, Ishikawa J, Matsuyama A, Ouchi N, Kihara S, Funahashi T, Tenner AJ, Tomiyama Y, Matsuzawa Y. Adiponectin, a new member of the family of soluble defense collagens, negatively regulates the growth of myelomonocytic progenitors and the functions of macrophages. Blood. 2000 Sep 1;96(5):1723-32. PMID 10961870
- [Background] Ouchi N, Kihara S, Arita Y, Nishida M, Matsuyama A, Okamoto Y, Ishigami M, Kuriyama H, Kishida K, Nishizawa H, Hotta K, Muraguchi M, Ohmoto Y, Yamashita S, Funahashi T, Matsuzawa Y. Adipocyte-derived plasma protein, adiponectin, suppresses lipid accumulation and class A scavenger receptor expression in human monocyte-derived macrophages. Circulation. 2001 Feb 27;103(8):1057-63. doi: 10.1161/01.cir.103.8.1057. PMID 11222466
- [Background] Miyazaki T, Shimada K, Mokuno H, Daida H. Adipocyte derived plasma protein, adiponectin, is associated with smoking status in patients with coronary artery disease. Heart. 2003 Jun;89(6):663. doi: 10.1136/heart.89.6.663. No abstract available. PMID 12748229
- [Background] Shimada K, Miyazaki T, Daida H. Adiponectin and atherosclerotic disease. Clin Chim Acta. 2004 Jun;344(1-2):1-12. doi: 10.1016/j.cccn.2004.02.020. PMID 15149866
- [Background] Matsuda M, Shimomura I, Sata M, Arita Y, Nishida M, Maeda N, Kumada M, Okamoto Y, Nagaretani H, Nishizawa H, Kishida K, Komuro R, Ouchi N, Kihara S, Nagai R, Funahashi T, Matsuzawa Y. Role of adiponectin in preventing vascular stenosis. The missing link of adipo-vascular axis. J Biol Chem. 2002 Oct 4;277(40):37487-91. doi: 10.1074/jbc.M206083200. Epub 2002 Jul 22. PMID 12138120
- [Background] Okamoto Y, Kihara S, Ouchi N, Nishida M, Arita Y, Kumada M, Ohashi K, Sakai N, Shimomura I, Kobayashi H, Terasaka N, Inaba T, Funahashi T, Matsuzawa Y. Adiponectin reduces atherosclerosis in apolipoprotein E-deficient mice. Circulation. 2002 Nov 26;106(22):2767-70. doi: 10.1161/01.cir.0000042707.50032.19. PMID 12451000
- [Background] Yamauchi T, Kamon J, Waki H, Imai Y, Shimozawa N, Hioki K, Uchida S, Ito Y, Takakuwa K, Matsui J, Takata M, Eto K, Terauchi Y, Komeda K, Tsunoda M, Murakami K, Ohnishi Y, Naitoh T, Yamamura K, Ueyama Y, Froguel P, Kimura S, Nagai R, Kadowaki T. Globular adiponectin protected ob/ob mice from diabetes and ApoE-deficient mice from atherosclerosis. J Biol Chem. 2003 Jan 24;278(4):2461-8. doi: 10.1074/jbc.M209033200. Epub 2002 Nov 12. PMID 12431986
- [Background] Kumada M, Kihara S, Sumitsuji S, Kawamoto T, Matsumoto S, Ouchi N, Arita Y, Okamoto Y, Shimomura I, Hiraoka H, Nakamura T, Funahashi T, Matsuzawa Y; Osaka CAD Study Group. Coronary artery disease. Association of hypoadiponectinemia with coronary artery disease in men. Arterioscler Thromb Vasc Biol. 2003 Jan 1;23(1):85-9. doi: 10.1161/01.atv.0000048856.22331.50. PMID 12524229
- [Background] Kojima S, Funahashi T, Sakamoto T, Miyamoto S, Soejima H, Hokamaki J, Kajiwara I, Sugiyama S, Yoshimura M, Fujimoto K, Miyao Y, Suefuji H, Kitagawa A, Ouchi N, Kihara S, Matsuzawa Y, Ogawa H. The variation of plasma concentrations of a novel, adipocyte derived protein, adiponectin, in patients with acute myocardial infarction. Heart. 2003 Jun;89(6):667. doi: 10.1136/heart.89.6.667. No abstract available. PMID 12748233
- [Background] Nakamura Y, Shimada K, Fukuda D, Shimada Y, Ehara S, Hirose M, Kataoka T, Kamimori K, Shimodozono S, Kobayashi Y, Yoshiyama M, Takeuchi K, Yoshikawa J. Implications of plasma concentrations of adiponectin in patients with coronary artery disease. Heart. 2004 May;90(5):528-33. doi: 10.1136/hrt.2003.011114. PMID 15084551
- [Background] Iwashima Y, Horio T, Suzuki Y, Kihara S, Rakugi H, Kangawa K, Funahashi T, Ogihara T, Kawano Y. Adiponectin and inflammatory markers in peripheral arterial occlusive disease. Atherosclerosis. 2006 Oct;188(2):384-90. doi: 10.1016/j.atherosclerosis.2005.10.039. PMID 16321391